CLINICAL TRIAL: NCT00818415
Title: An Open Label, Randomised Two Way Crossover Trial to Determine the Pharmacokinetic Profile of an Extended Release Naproxen Sodium Tablet Relative to Aleve Tablets Following Single and Multiple Dose Administration Under Fed Conditions.
Brief Title: Naproxen Sodium ER Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13965
Record Dates: First submitted 2008-12-08; First posted 2009-01-07 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Naproxen sodium ER (BAYH6689)
- Arm 2 (Active Comparator)
  Interventions: Drug: Commercial Naproxen (Aleve, BAYH6689)

INTERVENTIONS:
Drug: Naproxen sodium ER (BAYH6689) — Extented release Naproxen sodium (660mg) administered once a day
  Arms: Arm 1
Drug: Commercial Naproxen (Aleve, BAYH6689) — Immediate release Commercial Aleve (220mg) administered in a two ( 440 mg) plus one (220mg) dosing regime, 660 mg daily
  Arms: Arm 2

SUMMARY:
To determine the pharmacokinetic profile of the investigational product following dosing under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory, male and female volunteers between 18-55 years of age with a Body Mass Index (BMI) of approximately 18 to 30kg/m2, and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the principal Investigator and the Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g oral or patch contraceptives, intrauterine device, NuvaRing, Depo-Provera, or double-barrier and have a negative pregnancy test at Screening and Day 0 of each Dosing Period. Female subjects of non childbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy
* Be willing and able to participate in all scheduled visits, treatment plan, laboratory tests and other trial procedures according to the protocol
* Provide a personally signed and dated informed consent indicating that the subject has been informed of all pertinent aspects of the trial

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), naproxen sodium, or acetaminophen, and similar pharmacological agents or components of the products
* History of gastrointestinal bleeding or perforation, related to previous nonsteroidal anti-inflammatory drug (NSAID) therapy. Active, or history of recurrent peptic ulcer/ hemorrhage (two or more distinct episodes of proven ulceration or bleeding)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases or malignancies
* Have taken ASA, ASA-containing products, acetaminophen (acetyl-para-amino-phenol or APAP) or any other NSAID (Over the counter (OTC) or prescription) 7 days prior to dosing or during the treatment period, other than trial treatment
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product (e.g., nicotine patch, nicotine gum)
* Have taken any vitamin or herbal supplement within 7 days prior to dosing or refuse to refrain from use during the trial
* Alcoholism or drug abuse within 2 years prior to the Screening Visit
* Participation in any other trials involving investigational or marketed products within 30 days prior to the Screening Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) Profile of an extended release tablet of Naproxen Sodium under fed conditions | 4 weeks

SECONDARY OUTCOMES:
Assess the safety and tolerability of an extended release tablet of Naproxen Sodium | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Austin, Texas, United States